CLINICAL TRIAL: NCT03471936
Title: Right Ventricular Diastolic Function in Chronic Adverse RV Loading And Congenital Heart Disease
Acronym: RaDICAL-CHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator M.D. Ph. D. Philipp Lurz, Heart Center Leipzig - University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RADICAL001
Record Dates: First submitted 2018-02-01; First posted 2018-03-21 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Pulmonary Regurgitation; Congenital Heart Disease
Keywords: Congenital Heart Disease; pressure-volume loops; diastolic function
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Acquisition of pressure-volume loops (Other)
  Interventions: Diagnostic Test: Acquisition of pressure-volume-loops

INTERVENTIONS:
Diagnostic Test: Acquisition of pressure-volume-loops — Diagnostic workup including cardiac MRI, Echocardiography and cardiopulmonary exercise test (CPET) followed by invasive acquisition of RV and left ventricular (LV) pressure-volume-loops

SUMMARY:
The aim of the study is to assess the characteristics, incidence and predictors of load-independent right ventricle (RV) diastolic dysfunction in patients with congenital heart disease (CHD) and adverse RV loading conditions by acquiring pressure-volume loops and compare these results to a population of patients with exclusion of coronary artery disease and absence of any known disease affecting the RV.

DETAILED DESCRIPTION:
One of the major problems in the expanding population of patients with congenital heart disease (CHD) is dysfunction of the right ventricular (RV) outflow tract (OT). Initial surgical repair for complex conditions or repeated surgery for free pulmonary regurgitation often includes the creation of an artificial RV to main pulmonary artery connection. Over time, these conduits are prone to develop valvar incompetence or obstruction. There is clear evidence that pulmonary stenosis and pulmonary regurgitation are associated with exercise intolerance, arrhythmias and an increased risk of sudden death. Timely pulmonary valve replacement can halt and may reverse such unfavourable outcomes. However, this means that patients have to undergo multiple open-heart surgeries in order to reduce the haemodynamic burden on the right ventricle. Decision making in these patients with RVOT dysfunction is based on the aim to perform pulmonary valve replacement as late as possible to minimise the total number of open-heart surgeries required in individual patients, but before functional impairment might be irreversible. Importantly, this point of 'no return' in right ventricular pressure and/or volume overload is still unknown and represents one of the most challenging problems in the field of CHD. Ideally, quality of life, survival and freedom from atrial and ventricular arrhythmia should be the endpoints for any study trying to optimise timing of pulmonary valve replacement. However, such studies would require long follow-up in large patient populations and will not help to improve management of right ventricular outflow tract (RVOT) dysfunction in the short-term. In order to design studies with surrogate functional endpoints, a sound understanding of physiological consequences of altering RV loading and its implications for bi-ventricular function or exercise capacity is pivotal.

The investigators established a method of acquiring robust RV pressure-volume-loops at our institution. In the context of a research study, the investigators performed RV conductance catheter measurements in 22 patients with heart failure with preserved ejection fraction and in 11 patients with no evidence of any RV disease. Within the RaDICAL study the investigators aim further to compare these results to pressure-volume loops acquired in patients with congenital heart disease (CHD) and adverse RV loading conditions in order to evaluate characteristics, incidence and predictors of load-independent right ventricle (RV) diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CHD involving the RV
* Chronic RV volume and/or pressure overload as defined by:
* more than mild pulmonary regurgitation and/or
* more than mild tricuspid regurgitation and/or
* a gradient across the RV outflow tract of ≥ 3 m/s on echocardiography and/or
* estimated RV systolic pressure > 65 mmHg
* Clinical indication for cardiac catheterization
* Age 12 to 80 years
* Informed consent

Exclusion Criteria:

* Contraindication for magnetic resonance imaging or cardiopulmonary exercise testing
* Pregnancy
* RV systolic function on magnetic resonance imaging < 45%

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07-07 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Presence of RV diastolic dysfunction in CHD and RVOT dysfunction | Baseline
  Determination of load-independent stiffness constant in CHD

SECONDARY OUTCOMES:
Link between RV load-independent stiffness constant and functional capacity | Baseline
  Oxygen uptake (VO2 max) in correlation to load-independent stiffness constant
Association between E/É and RV stiffness in CHD | Baseline
  Correlation between E/É and load-independent stiffness constant
Association between RV stiffness expressed as E/É and functional outcome after surgical or percutaneous pulmonary valve replacement | 6 months
  Correlation between E/É before intervention and VO2 max change after pulmonary valve replacement

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Dähnert, MD, Principal Investigator — Head of pediatric cardiology, Heart Center Leipzig
Locations (1):
- Heart Center of the University Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown JW, Ruzmetov M, Rodefeld MD, Vijay P, Turrentine MW. Right ventricular outflow tract reconstruction with an allograft conduit in non-ross patients: risk factors for allograft dysfunction and failure. Ann Thorac Surg. 2005 Aug;80(2):655-63; discussion 663-4. doi: 10.1016/j.athoracsur.2005.02.053. PMID 16039222
- [Background] Rastan AJ, Walther T, Daehnert I, Hambsch J, Mohr FW, Janousek J, Kostelka M. Bovine jugular vein conduit for right ventricular outflow tract reconstruction: evaluation of risk factors for mid-term outcome. Ann Thorac Surg. 2006 Oct;82(4):1308-15. doi: 10.1016/j.athoracsur.2006.04.071. PMID 16996925
- [Background] Stark J, Bull C, Stajevic M, Jothi M, Elliott M, de Leval M. Fate of subpulmonary homograft conduits: determinants of late homograft failure. J Thorac Cardiovasc Surg. 1998 Mar;115(3):506-14; discussion 514-6. doi: 10.1016/S0022-5223(98)70312-5. PMID 9535436
- [Background] Tweddell JS, Pelech AN, Frommelt PC, Mussatto KA, Wyman JD, Fedderly RT, Berger S, Frommelt MA, Lewis DA, Friedberg DZ, Thomas JP Jr, Sachdeva R, Litwin SB. Factors affecting longevity of homograft valves used in right ventricular outflow tract reconstruction for congenital heart disease. Circulation. 2000 Nov 7;102(19 Suppl 3):III130-5. doi: 10.1161/01.cir.102.suppl_3.iii-130. PMID 11082375
- [Background] Gatzoulis MA, Balaji S, Webber SA, Siu SC, Hokanson JS, Poile C, Rosenthal M, Nakazawa M, Moller JH, Gillette PC, Webb GD, Redington AN. Risk factors for arrhythmia and sudden cardiac death late after repair of tetralogy of Fallot: a multicentre study. Lancet. 2000 Sep 16;356(9234):975-81. doi: 10.1016/S0140-6736(00)02714-8. PMID 11041398
- [Background] Carvalho JS, Shinebourne EA, Busst C, Rigby ML, Redington AN. Exercise capacity after complete repair of tetralogy of Fallot: deleterious effects of residual pulmonary regurgitation. Br Heart J. 1992 Jun;67(6):470-3. doi: 10.1136/hrt.67.6.470. PMID 1622697
- [Background] Lurz P, Puranik R, Nordmeyer J, Muthurangu V, Hansen MS, Schievano S, Marek J, Bonhoeffer P, Taylor AM. Improvement in left ventricular filling properties after relief of right ventricle to pulmonary artery conduit obstruction: contribution of septal motion and interventricular mechanical delay. Eur Heart J. 2009 Sep;30(18):2266-74. doi: 10.1093/eurheartj/ehp258. Epub 2009 Jun 26. PMID 19561027
- [Background] Lurz P, Riede FT, Taylor AM, Wagner R, Nordmeyer J, Khambadkone S, Kinzel P, Derrick G, Schuler G, Bonhoeffer P, Giardini A, Daehnert I. Impact of percutaneous pulmonary valve implantation for right ventricular outflow tract dysfunction on exercise recovery kinetics. Int J Cardiol. 2014 Nov 15;177(1):276-80. doi: 10.1016/j.ijcard.2014.09.014. Epub 2014 Sep 22. PMID 25499392
- [Background] Lurz P, Nordmeyer J, Muthurangu V, Khambadkone S, Derrick G, Yates R, Sury M, Bonhoeffer P, Taylor AM. Comparison of bare metal stenting and percutaneous pulmonary valve implantation for treatment of right ventricular outflow tract obstruction: use of an x-ray/magnetic resonance hybrid laboratory for acute physiological assessment. Circulation. 2009 Jun 16;119(23):2995-3001. doi: 10.1161/CIRCULATIONAHA.108.836312. Epub 2009 Jun 1. PMID 19487596
- [Background] Lurz P, Coats L, Khambadkone S, Nordmeyer J, Boudjemline Y, Schievano S, Muthurangu V, Lee TY, Parenzan G, Derrick G, Cullen S, Walker F, Tsang V, Deanfield J, Taylor AM, Bonhoeffer P. Percutaneous pulmonary valve implantation: impact of evolving technology and learning curve on clinical outcome. Circulation. 2008 Apr 15;117(15):1964-72. doi: 10.1161/CIRCULATIONAHA.107.735779. Epub 2008 Apr 7. PMID 18391109
- [Background] Burkhoff D, Mirsky I, Suga H. Assessment of systolic and diastolic ventricular properties via pressure-volume analysis: a guide for clinical, translational, and basic researchers. Am J Physiol Heart Circ Physiol. 2005 Aug;289(2):H501-12. doi: 10.1152/ajpheart.00138.2005. PMID 16014610
- [Background] Dimopoulos K, Okonko DO, Diller GP, Broberg CS, Salukhe TV, Babu-Narayan SV, Li W, Uebing A, Bayne S, Wensel R, Piepoli MF, Poole-Wilson PA, Francis DP, Gatzoulis MA. Abnormal ventilatory response to exercise in adults with congenital heart disease relates to cyanosis and predicts survival. Circulation. 2006 Jun 20;113(24):2796-802. doi: 10.1161/CIRCULATIONAHA.105.594218. Epub 2006 Jun 12. PMID 16769913